CLINICAL TRIAL: NCT03706885
Title: A Proof-of-Concept Clinical Research Study of Efavirenz in Patients With Alzheimer's Disease
Brief Title: Efavirenz for Patients With Alzheimer's Disease
Acronym: EPAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Irina Pikuleva, PhD, Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ADDF 20160601
Record Dates: First submitted 2018-08-15; First posted 2018-10-16 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease | interventions — efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the Statistician and Pharmacists are unmasked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Treatment with placebo - 1 pill per day for 20 weeks
  Interventions: Drug: Sustiva Pill
- Sustiva 50mg (Active Comparator): Treatment with Sustiva 50mg - 1 pill per day for 20 weeks
  Interventions: Drug: Sustiva Pill
- Sustiva 200mg (Active Comparator): Treatment with Sustiva 200mg - 1 pill per day for 20 weeks
  Interventions: Drug: Sustiva Pill

INTERVENTIONS:
Drug: Sustiva Pill — One pill (Sustiva 50 mg or Sustiva 200mg or Placebo) One pill per day for 20 weeks
  Other Names: Efavirenz

SUMMARY:
This will be a two-center, placebo controlled blinded clinical trial to evaluate the safety and tolerability of efavirenz (EFV) in 36 clinically stable subjects with mild cognitive impairment/early dementia due to Alzheimer's Disease (AD) age ≥55 years. Of these 36 total subjects, 18 will be recruited by MGH and 18 will be recruited by UH. A subset of the subjects at MGH only will also participate in a Stable Isotope Labeling Kinetics (SILK) protocol with deuterated water (a nonhazardous substance), designed to more precisely measure EFV effects on CNS cholesterol turnover.

Each respective site's 18 total recruited individuals will be divided into 3 groups: these 3 groups will represent two particular dosages of EFV and a placebo group, respectively. In a double-blind fashion, participants will be receiving either a capsule of EFV or placebo daily for 20 weeks. At MGH only, 12 individuals (4 from each of the two EFV groups and placebo) will participate in the unique "heavy water" SILK protocol assessing the kinetics of deuterium enrichment in plasma 24-hydroxycholesterol (24-OHC). All study participants at both sites will have their blood, cerebral spinal fluid, and urine analyzed at various points throughout the study. All participants will have their DNA genotyped for APOE isoforms (E2, E3 or E4) and single nucleotide polymorphisms (SNPs) in CYP46A1 (rs754203) and CYP2B6 (rs3745274) to be used for post-hoc analysis.

DETAILED DESCRIPTION:
1.0 BACKGROUND

1.1. Introduction

The brain is the most cholesterol-rich organ in the body. Circulating peripheral cholesterol cannot cross the blood-brain barrier and enter the brain, so all of cerebral cholesterol is synthesized and metabolized locally. The CNS relies on cholesterol 24-hydroxylation as its major mechanism for eliminating excess cholesterol from the brain. CYP46A1 is an enzyme of the CNS responsible for hydroxylating cholesterol to 24-hydroxycholesterol (24-OHC), which can easily pass the blood-brain barrier and leave the brain to travel into the systemic blood circulation. In fact, 24-OHC plasma level is a specific biomarker for cholesterol homeostasis and CYP46A1 activity in the brain. 24-OHC is a potent modulator of NMDAR, a receptor system in the brain whose hypofunctioning can lead to problems of memory and learning performance. Cyp46a1-/- mice and CYP46A1 transgenic animals established that CYP46A1 is involved in higher-order brain functions and processes beyond mere cholesterol balance: the Cyp46a1-/- mice lacking CYP46A1 demonstrated severe deficiencies in spatial, associative, and motor learning-- as well as deficiencies in long-term potentiation of the hippocampus. On the other hand, CYP46A1 transgenic animals with an abundance of CYP46A1 had improvements in spatial memory and significant increase in the levels of NMDAR in the hippocampus. CYP46A1 overexpressing mice possessing an animal model of AD demonstrated improvements in learning and memory, and reduction in pathological amyloid beta.

Various studies have demonstrated a number of associations between CYP46A1 and AD. For unknown reasons, this neuron-specific enzyme becomes specifically expressed in astrocytes of AD patients; plasma levels of 24-OHC, the product of CYP46A1, also change in AD patients-there are slight elevations of plasma levels in the early stages of AD, followed by decreases in the later stages of AD, (the elevations have been interpreted to represent demyelination of the brain and subsequent release of 24-OHC into the systemic circulation, and the decreases could be attributed to loss of CYP46A1 during the physical process of neuronal degeneration); and, finally, CYP46A1 is highly polymorphic enzyme with the most frequent intronic SNPs (rs754203, rs3742376, rs7157609, and rs4900442 being found at ~29- 40% frequency in the population. The CYP46A1-AD genetic link is, however, unclear, with only about half of linkage studies establishing the CYP46A1-AD association. Data from several laboratories point to enhanced metabolism of cerebral cholesterol as a strong anti-AD disease mechanism.

CYP46A1-mediated metabolism of cerebral cholesterol has never been considered as a pharmacologic target because the proposed activity requires activation of the enzyme, a significant challenge for drug developers. Only 5% of drugs on the market act as enzyme activators, with the majority of pharmaceuticals serving as enzyme inhibitors. Dr. Pikuleva's laboratory--over the course of more than 10 years' work--overcame this challenge by ultimately discovering that in mice, CYP46A1 can indeed be activated pharmacologically by efavirenz (EFV). This CYP46A1 activation also leads to enhanced cerebral cholesterol turnover in mice.

2.0 STUDY RATIONALE

AD has been shown to be a disease featuring rampant aberrant cerebral cholesterol phenomenon; hence the AD population is the most appropriate demographic to include in this study. The investigators expect EFV to be a cerebral cholesterol-metabolism-modifying medication, which may have prolific uses in neurodegenerative diseases--such as AD--where cholesterol metabolism is aberrant.

2.1. Risk/Benefit Assessment

EFV is an FDA-approved anti-retroviral medication for use in the adult population-including the geriatric population. The current recommended dose of Sustiva for adults with HIV is 600 mg daily. This research study will be utilizing very low doses of Sustiva (50 mg and 200 mg), which are the current dosage ranges for children. The investigators have no reason to believe that utilizing 1/3 the adult dose of a drug in the geriatric population will increase the risk of the drug beyond those side effects which are already listed for this product. The study participants will be monitored very closely throughout the course of the research study to bring to light any untoward effects in the participants that would outweigh the potential benefit of this study.

3.0 STUDY OBJECTIVES

3.1. Primary Objectives

* To ascertain if EFV engages CYP46A1 and affects brain cholesterol metabolism.
* To investigate whether EFV alters plasma 24-OHC concentrations.
* To confirm the safety and tolerability of low doses of EFV.

3.2. Secondary Objectives

● To precisely measure EFV's effect on CYP46A1 activation and CNS-cholesterol turnover via Stable Isotope Labeling Kinetics (SILK) study.

3.3. Tertiary Objectives

● To conduct post-hoc analysis to investigate whether APOE isorforms and SNPs in CYP46A1 and CYP2B6 affect study participant response to EFV.

4.0 STUDY DESIGN

4.1. Study Design Overview

A total of 36 patients will be enrolled at 2 sites, 18 patients at the UH site and 18 patients at the MGH site. Site UH, the recruiting clinician at this site is Alan Lerner, MD. Site MGH, recruiting clinician at this site is Steven Arnold, MD. At each site, subjects will be divided into 3 groups; Group1 will consist of 6 subjects who will receive 50 mg EFV; Group 2 will consist of 6 subjects who will receive 200 mg EFV and Group 3 will consist of 6 subjects who will receive Placebo.

5.0 CRITERIA FOR EVALUATIONS

5.1. Primary Endpoints

CYP46A1 engagement will be indicated either by a decrease or increase in plasma 24-OHC from baseline to final time of treatment in the study participants receiving EFV.

CYP46A1 activation will be indicated by ≥ 30% increase in plasma 24-OHC from baseline to final time of treatment in the study participants receiving EFV. The primary dose selection criterion for EFV will be to maximize the proportion of subjects that exceed the threshold for 24-OHC increase, provided there are no associated safety concerns.

A "symptom checklist" will be reviewed and asked of the study participants every two weeks to ensure that no untoward, serious complications arise from treatment with EFV. It is not expected that any serious adverse events will occur. All participants will conclude their treatment with a Post-Study Safety Check Visit during Week 22.

5.2. Secondary Endpoints

Plasma levels of deuterated 24-OHC in patients involved in the SILK study, who will drink deuterated water, will be measured to evaluate EFV's effect on CNS-cholesterol turnover.

5.3. Tertiary Endpoints

Carriers of the APOE E4 allele could be better responders to the anti-AD effects of EFV because in the brain, cholesterol output is a function of both APOE-mediated cholesterol transport and CYP46A1-mediated cholesterol metabolism. Accordingly, if one of these pathways is impaired, like in APOE E4 carriers, the significance of the other pathway is increased. Similarly, the CYP46A1 polymorphisms may affect the ability of EFV to increase 24-OHC because the baseline levels of CYP46A1 and 24-OHC in the carriers of these polymorphisms could be lower, if these polymorphisms affect CYP46A1 protein levels. Finally, at a high dose (400-600 mg/day), plasma concentrations of EFV depend on the frequent SNP rs3745274 in CYP2B6 that metabolizes EFV. Genotyping will be carried out by the Molecular Biology and Genotyping Module at Case Western Reserve University.

6.0 SUBJECT SELECTION

A total of 36 participants, either male or female, will be enrolled between the ages of 55-85 for 22 weeks. Recruitment of study participants will occur during potential participants' regularly-schedule clinical visits, or from chart review.

6.1. Study Population

All participants should have either mild cognitive impairment or early dementia due to AD, defined clinically as follows:

* Complaint of cognitive decline
* Mini-Mental Status Examination (MMSE) totaling between 16-30
* Clinical Dementia Rating (CDR) equaling 0.5-1

The 36 study participants will be recruited in a timeframe of approximately 8-9 months. The two study sites are anticipated to recruit 2 study participants per month. This anticipated rate is based on the investigators previous experience in clinical study subject enrollment and high patient volume at the University Hospitals Brain Health and Memory Center and the Memory Disorders Clinic, and the Memory Disorders Unit and Massachusetts Alzheimer's Disease Research Center (MADRC) at Massachusetts General Hospitals (MGH).

7.0 CONCOMITANT THERAPIES

Medical history will be collected for all medications at the screening visit and at all subsequent clinical and telephone follow-up visits. All subjects should be maintained on the same medications from screening through Visit 7, as medically feasible, with no introduction of new therapies.If any changes in concomitant medications are made for any reason by the study participant's personal physician(s), the changes and reason(s) for the change(s) will be documented.

7.1. Allowed

Except as noted in the prohibited medications section 7.2. Stable use of cholinesterase inhibitor is permitted if doses are stable for 3 months prior to enrollment.

7.2. Prohibited

EFV is mainly metabolized by CYP2B6 and CYP3A4, and in the 600 mg/day dose range or higher, has potential interactions with other drugs. EFV is expected to stimulate cholesterol elimination from the brain, inducing a compensatory upregulation of cerebral cholesterol biosynthesis; statins that cross the blood-brain barrier would be expected to especially inhibit cerebral cholesterol biosynthesis and confound 24-OHC biomarking of EFV's effect. Study participants in the clinical research study should not have taken the following medication within 3 months of commencing their participatory role in the study: simvastatin, antiepileptic agents, clopidogrel, voriconazole, systemic ketoconazole, cyclosporine, St. John's Wort.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 55-85
* Either male or female
* Diagnosis of (a) as per below:

  a) Mild Cognitive Impairment (MCI) or early dementia due to AD as defined by (1) complaint of cognitive decline, (2) MMSE Total=16-30, (3) CDR=0.5-1
* Fluent in English
* Education >8 years, literate, and/or good working history that precludes consideration of mental retardation
* Visual and auditory acuity sufficient for neuropsychological testing
* Modified Hachinski Ischemic Score<4
* No major health issues or diseases expected to interfere with the study
* Willing to complete all assessments and study procedures
* Not pregnant, lactating or of child-bearing potential (women must be >2 years post- menopausal or surgically sterile)
* If cognitively impaired, study partner with frequent contact with patient willing to accompany patient to visits and complete partner study forms
* No contraindication or hypersensitivity to EFV
* Screening laboratory testing must be within normal limits or, if abnormal, must be judged to be clinically insignificant by the investigators
* Stable use of cholinesterase inhibitor is permitted if doses are stable for 3 months prior to enrollment

Exclusion Criteria:

* Any CNS disease other than suspected prodromal or early AD, such as clinical stroke, brain tumor, normal pressure hydrocephalus, brain tumor, multiple sclerosis, significant head trauma with persistent neurological or cognitive deficits or complaints, Parkinson's Disease, frontotemporal dementia, or other neurodegenerative diseases
* Ongoing major and active psychiatric disorder and/or other concurrent medical condition that, in the opinion of the investigator, might compromise safety and/or compliance with study requirements.
* History of alcohol or other substance abuse or dependence within the past two years
* Any significant systemic illness or unstable medical condition that could affect study compliance, including a history of prolonged QTc
* Laboratory abnormalities in B12, TSH, or other common laboratory parameters that might contribute to cognitive dysfunction
* Current use of medications with psychoactive properties that may deleteriously affect cognition (e.g., anticholinergics, antihistamines, antipsychotics, sedative hypnotics, anxiolytics) that, in the opinion of the investigator, may deleteriously affect cognition. Use of other investigational agents one month prior to entry and for the duration of the study
* Treatment with any of the following agents/classes within the past 3 months: simvastatin, antiepileptic agents, clopidogrel, voriconazole, systemic ketoconazole, cyclosporine, St. John's Wort.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Plasma levels of 24-hydroxycholesterol | 1 year
  Changes in plasma 24-hydroxycholesterol (measured in ng/dL) by more or equal to 30%.

SECONDARY OUTCOMES:
Plasma levels of deuterated 24-hydroxycholesterol | 1 year
  Plasma appearance of deuterated 24-hydroxycholetserol (measured in ng/dL) will be measured within 14 days after a participant will drink the last portion of deuterated water in the Stable Isotope Kinetics Labeling Study.
APOE isoform status (E2, E3, or E4) and presence of the SNPs rs754203 and rs3745274 in CYP46A1 and CYP2B6, respectively. | 1 year
  Participants will be genotyped for the APOE isoform status (E2, E3, or E4) and presence of the SNPs rs754203 and rs3745274 in CYP46A1 and CYP2B6, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Irina A Pikuleva, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Brain Health and Memory Center, Beachwood, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dietschy JM, Turley SD. Thematic review series: brain Lipids. Cholesterol metabolism in the central nervous system during early development and in the mature animal. J Lipid Res. 2004 Aug;45(8):1375-97. doi: 10.1194/jlr.R400004-JLR200. PMID 15254070
- [Background] Lutjohann D, Breuer O, Ahlborg G, Nennesmo I, Siden A, Diczfalusy U, Bjorkhem I. Cholesterol homeostasis in human brain: evidence for an age-dependent flux of 24S-hydroxycholesterol from the brain into the circulation. Proc Natl Acad Sci U S A. 1996 Sep 3;93(18):9799-804. doi: 10.1073/pnas.93.18.9799. PMID 8790411
- [Background] Lund EG, Xie C, Kotti T, Turley SD, Dietschy JM, Russell DW. Knockout of the cholesterol 24-hydroxylase gene in mice reveals a brain-specific mechanism of cholesterol turnover. J Biol Chem. 2003 Jun 20;278(25):22980-8. doi: 10.1074/jbc.M303415200. Epub 2003 Apr 9. PMID 12686551
- [Background] Lund EG, Guileyardo JM, Russell DW. cDNA cloning of cholesterol 24-hydroxylase, a mediator of cholesterol homeostasis in the brain. Proc Natl Acad Sci U S A. 1999 Jun 22;96(13):7238-43. doi: 10.1073/pnas.96.13.7238. PMID 10377398
- [Background] Ramirez DM, Andersson S, Russell DW. Neuronal expression and subcellular localization of cholesterol 24-hydroxylase in the mouse brain. J Comp Neurol. 2008 Apr 10;507(5):1676-93. doi: 10.1002/cne.21605. PMID 18241055
- [Background] Meaney S, Bodin K, Diczfalusy U, Bjorkhem I. On the rate of translocation in vitro and kinetics in vivo of the major oxysterols in human circulation: critical importance of the position of the oxygen function. J Lipid Res. 2002 Dec;43(12):2130-5. doi: 10.1194/jlr.m200293-jlr200. PMID 12454275
- [Background] Leoni V, Caccia C. 24S-hydroxycholesterol in plasma: a marker of cholesterol turnover in neurodegenerative diseases. Biochimie. 2013 Mar;95(3):595-612. doi: 10.1016/j.biochi.2012.09.025. Epub 2012 Oct 3. PMID 23041502
- [Background] Bretillon L, Lutjohann D, Stahle L, Widhe T, Bindl L, Eggertsen G, Diczfalusy U, Bjorkhem I. Plasma levels of 24S-hydroxycholesterol reflect the balance between cerebral production and hepatic metabolism and are inversely related to body surface. J Lipid Res. 2000 May;41(5):840-5. PMID 10787445
- [Background] Paul SM, Doherty JJ, Robichaud AJ, Belfort GM, Chow BY, Hammond RS, Crawford DC, Linsenbardt AJ, Shu HJ, Izumi Y, Mennerick SJ, Zorumski CF. The major brain cholesterol metabolite 24(S)-hydroxycholesterol is a potent allosteric modulator of N-methyl-D-aspartate receptors. J Neurosci. 2013 Oct 30;33(44):17290-300. doi: 10.1523/JNEUROSCI.2619-13.2013. PMID 24174662
- [Background] Kotti TJ, Ramirez DM, Pfeiffer BE, Huber KM, Russell DW. Brain cholesterol turnover required for geranylgeraniol production and learning in mice. Proc Natl Acad Sci U S A. 2006 Mar 7;103(10):3869-74. doi: 10.1073/pnas.0600316103. Epub 2006 Feb 27. PMID 16505352
- [Background] Maioli S, Bavner A, Ali Z, Heverin M, Ismail MA, Puerta E, Olin M, Saeed A, Shafaati M, Parini P, Cedazo-Minguez A, Bjorkhem I. Is it possible to improve memory function by upregulation of the cholesterol 24S-hydroxylase (CYP46A1) in the brain? PLoS One. 2013 Jul 16;8(7):e68534. doi: 10.1371/journal.pone.0068534. Print 2013. PMID 23874659
- [Background] Hudry E, Van Dam D, Kulik W, De Deyn PP, Stet FS, Ahouansou O, Benraiss A, Delacourte A, Bougneres P, Aubourg P, Cartier N. Adeno-associated virus gene therapy with cholesterol 24-hydroxylase reduces the amyloid pathology before or after the onset of amyloid plaques in mouse models of Alzheimer's disease. Mol Ther. 2010 Jan;18(1):44-53. doi: 10.1038/mt.2009.175. Epub 2009 Aug 4. PMID 19654569
- [Background] Bryleva EY, Rogers MA, Chang CC, Buen F, Harris BT, Rousselet E, Seidah NG, Oddo S, LaFerla FM, Spencer TA, Hickey WF, Chang TY. ACAT1 gene ablation increases 24(S)-hydroxycholesterol content in the brain and ameliorates amyloid pathology in mice with AD. Proc Natl Acad Sci U S A. 2010 Feb 16;107(7):3081-6. doi: 10.1073/pnas.0913828107. Epub 2010 Jan 26. PMID 20133765
- [Background] Bogdanovic N, Bretillon L, Lund EG, Diczfalusy U, Lannfelt L, Winblad B, Russell DW, Bjorkhem I. On the turnover of brain cholesterol in patients with Alzheimer's disease. Abnormal induction of the cholesterol-catabolic enzyme CYP46 in glial cells. Neurosci Lett. 2001 Nov 13;314(1-2):45-8. doi: 10.1016/s0304-3940(01)02277-7. PMID 11698143
- [Background] Radhakrishnan A, Sun LP, Kwon HJ, Brown MS, Goldstein JL. Direct binding of cholesterol to the purified membrane region of SCAP: mechanism for a sterol-sensing domain. Mol Cell. 2004 Jul 23;15(2):259-68. doi: 10.1016/j.molcel.2004.06.019. PMID 15260976
- [Background] Lutjohann D, Papassotiropoulos A, Bjorkhem I, Locatelli S, Bagli M, Oehring RD, Schlegel U, Jessen F, Rao ML, von Bergmann K, Heun R. Plasma 24S-hydroxycholesterol (cerebrosterol) is increased in Alzheimer and vascular demented patients. J Lipid Res. 2000 Feb;41(2):195-8. PMID 10681402
- [Background] Russell DW, Halford RW, Ramirez DM, Shah R, Kotti T. Cholesterol 24-hydroxylase: an enzyme of cholesterol turnover in the brain. Annu Rev Biochem. 2009;78:1017-40. doi: 10.1146/annurev.biochem.78.072407.103859. PMID 19489738
- [Background] Mast N, Norcross R, Andersson U, Shou M, Nakayama K, Bjorkhem I, Pikuleva IA. Broad substrate specificity of human cytochrome P450 46A1 which initiates cholesterol degradation in the brain. Biochemistry. 2003 Dec 9;42(48):14284-92. doi: 10.1021/bi035512f. PMID 14640697
- [Background] Mast N, Andersson U, Nakayama K, Bjorkhem I, Pikuleva IA. Expression of human cytochrome P450 46A1 in Escherichia coli: effects of N- and C-terminal modifications. Arch Biochem Biophys. 2004 Aug 1;428(1):99-108. doi: 10.1016/j.abb.2004.05.012. PMID 15234274
- [Background] White MA, Mast N, Bjorkhem I, Johnson EF, Stout CD, Pikuleva IA. Use of complementary cation and anion heavy-atom salt derivatives to solve the structure of cytochrome P450 46A1. Acta Crystallogr D Biol Crystallogr. 2008 May;64(Pt 5):487-95. doi: 10.1107/S0907444908004046. Epub 2008 Apr 19. PMID 18453684
- [Background] Mast N, White MA, Bjorkhem I, Johnson EF, Stout CD, Pikuleva IA. Crystal structures of substrate-bound and substrate-free cytochrome P450 46A1, the principal cholesterol hydroxylase in the brain. Proc Natl Acad Sci U S A. 2008 Jul 15;105(28):9546-51. doi: 10.1073/pnas.0803717105. Epub 2008 Jul 9. PMID 18621681
- [Background] Mast N, Saadane A, Valencia-Olvera A, Constans J, Maxfield E, Arakawa H, Li Y, Landreth G, Pikuleva IA. Cholesterol-metabolizing enzyme cytochrome P450 46A1 as a pharmacologic target for Alzheimer's disease. Neuropharmacology. 2017 Sep 1;123:465-476. doi: 10.1016/j.neuropharm.2017.06.026. Epub 2017 Jun 24. PMID 28655608
- [Background] Liao WL, Dodder NG, Mast N, Pikuleva IA, Turko IV. Steroid and protein ligand binding to cytochrome P450 46A1 as assessed by hydrogen-deuterium exchange and mass spectrometry. Biochemistry. 2009 May 19;48(19):4150-8. doi: 10.1021/bi900168m. PMID 19317426
- [Background] Mast N, Liao WL, Pikuleva IA, Turko IV. Combined use of mass spectrometry and heterologous expression for identification of membrane-interacting peptides in cytochrome P450 46A1 and NADPH-cytochrome P450 oxidoreductase. Arch Biochem Biophys. 2009 Mar 1;483(1):81-9. doi: 10.1016/j.abb.2009.01.002. Epub 2009 Jan 10. PMID 19161969
- [Background] Mast N, Charvet C, Pikuleva IA, Stout CD. Structural basis of drug binding to CYP46A1, an enzyme that controls cholesterol turnover in the brain. J Biol Chem. 2010 Oct 8;285(41):31783-95. doi: 10.1074/jbc.M110.143313. Epub 2010 Jul 28. PMID 20667828
- [Background] Mast N, Linger M, Clark M, Wiseman J, Stout CD, Pikuleva IA. In silico and intuitive predictions of CYP46A1 inhibition by marketed drugs with subsequent enzyme crystallization in complex with fluvoxamine. Mol Pharmacol. 2012 Nov;82(5):824-34. doi: 10.1124/mol.112.080424. Epub 2012 Aug 2. PMID 22859721
- [Background] Mast N, Zheng W, Stout CD, Pikuleva IA. Binding of a cyano- and fluoro-containing drug bicalutamide to cytochrome P450 46A1: unusual features and spectral response. J Biol Chem. 2013 Feb 15;288(7):4613-24. doi: 10.1074/jbc.M112.438754. Epub 2013 Jan 3. PMID 23288837
- [Background] Mast N, Zheng W, Stout CD, Pikuleva IA. Antifungal Azoles: Structural Insights into Undesired Tight Binding to Cholesterol-Metabolizing CYP46A1. Mol Pharmacol. 2013 Jul;84(1):86-94. doi: 10.1124/mol.113.085902. Epub 2013 Apr 19. PMID 23604141
- [Background] Mast N, Li Y, Linger M, Clark M, Wiseman J, Pikuleva IA. Pharmacologic stimulation of cytochrome P450 46A1 and cerebral cholesterol turnover in mice. J Biol Chem. 2014 Feb 7;289(6):3529-38. doi: 10.1074/jbc.M113.532846. Epub 2013 Dec 18. PMID 24352658
- [Background] Fanara P, Wong PY, Husted KH, Liu S, Liu VM, Kohlstaedt LA, Riiff T, Protasio JC, Boban D, Killion S, Killian M, Epling L, Sinclair E, Peterson J, Price RW, Cabin DE, Nussbaum RL, Bruhmann J, Brandt R, Christine CW, Aminoff MJ, Hellerstein MK. Cerebrospinal fluid-based kinetic biomarkers of axonal transport in monitoring neurodegeneration. J Clin Invest. 2012 Sep;122(9):3159-69. doi: 10.1172/JCI64575. Epub 2012 Aug 27. PMID 22922254
- [Background] Lam TN, Hui KH, Chan DP, Lee SS. Genotype-guided dose adjustment for the use of efavirenz in HIV treatment. J Infect. 2015 Nov;71(5):607-9. doi: 10.1016/j.jinf.2015.07.005. Epub 2015 Jul 18. No abstract available. PMID 26196596
- [Background] Apostolova N, Funes HA, Blas-Garcia A, Galindo MJ, Alvarez A, Esplugues JV. Efavirenz and the CNS: what we already know and questions that need to be answered. J Antimicrob Chemother. 2015 Oct;70(10):2693-708. doi: 10.1093/jac/dkv183. Epub 2015 Jul 22. PMID 26203180
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] Hughes CP, Berg L, Danziger WL, Coben LA, Martin RL. A new clinical scale for the staging of dementia. Br J Psychiatry. 1982 Jun;140:566-72. doi: 10.1192/bjp.140.6.566. PMID 7104545
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Dzeletovic S, Breuer O, Lund E, Diczfalusy U. Determination of cholesterol oxidation products in human plasma by isotope dilution-mass spectrometry. Anal Biochem. 1995 Feb 10;225(1):73-80. doi: 10.1006/abio.1995.1110. PMID 7778789
- [Background] Mast N, Reem R, Bederman I, Huang S, DiPatre PL, Bjorkhem I, Pikuleva IA. Cholestenoic Acid is an important elimination product of cholesterol in the retina: comparison of retinal cholesterol metabolism with that in the brain. Invest Ophthalmol Vis Sci. 2011 Feb 1;52(1):594-603. doi: 10.1167/iovs.10-6021. Print 2011 Jan. PMID 20881306
- [Background] Kotti T, Head DD, McKenna CE, Russell DW. Biphasic requirement for geranylgeraniol in hippocampal long-term potentiation. Proc Natl Acad Sci U S A. 2008 Aug 12;105(32):11394-9. doi: 10.1073/pnas.0805556105. Epub 2008 Aug 6. PMID 18685105
- [Result] Lerner AJ, Arnold SE, Maxfield E, Koenig A, Toth ME, Fortin B, Mast N, Trombetta BA, Denker J, Pieper AA, Tatsuoka C, Raghupathy S, Pikuleva IA. CYP46A1 activation by low-dose efavirenz enhances brain cholesterol metabolism in subjects with early Alzheimer's disease. Alzheimers Res Ther. 2022 Dec 29;14(1):198. doi: 10.1186/s13195-022-01151-z. PMID 36581878
- [Derived] Gascon-Bayarri J, Simon PC, Llop R, Carnaval T, Ledesma MD, Rico I, Sanchez-Castaneda C, Campdelacreu-Fumado J, Calvo-Malvar N, Cos M, de Lama E, Cortes-Romera M, Rodriguez-Bel L, Perez-Sousa C, Cerdan Sanchez M, Muelas N, Sevillano MD, Mir P, Lopez de Munain A, Ferrer A, Videla S. Efficacy and safety clinical trial with efavirenz in patients diagnosed with adult Niemann-pick type C with cognitive impairment. Medicine (Baltimore). 2022 Dec 2;101(48):e31471. doi: 10.1097/MD.0000000000031471. PMID 36482560